CLINICAL TRIAL: NCT05962762
Title: A Clinical Trial to Evaluate the Safety, Tolerance and Efficacy of aCell Injection of Allogeneic UC-MSCs in Patients With Ankylosing Spondylitis
Brief Title: Safety and Tolerance of Umbilical Cord Mesenchymal Stem Cells (UC-MSC) in Patients With Ankylosing Spondylitis
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Asia Cell Therapeutics (Shanghai) Co., Ltd. (Industry)
Collaborators: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: QS-AS-S1
Record Dates: First submitted 2023-05-25; First posted 2023-07-27 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Ankylosing Spondylitis
Keywords: Human umbilical cord mesenchymal stem cell; ankylosing spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Human Umbilical Cord Mesenchymal Stem Cell Injection (Experimental): The trial was divided into three dose groups： Low-dose group: 1000000 cells/kg Medium-dose group: 3000000 cells/kg High-does group: 5000000 cells/kg
  Interventions: Biological: Human Umbilical Cord Mesenchymal Stem Cells

INTERVENTIONS:
Biological: Human Umbilical Cord Mesenchymal Stem Cells — The trial was conducted sequentially from the low dose group to the high dose group, with 3-6 subjects enrolled in each dose group. The trial was conducted on a case-by-case basis in the high dose group, with each subject in the high dose group being enrolled in subsequent subjects only after completion of at least 7 days of post-dose safety observation. Each subject received only one corresponding dose. All subjects received experimental drugs and conventional treatment during the study period.
  All subjects in each test dose group will complete a 4-week (28-day) dose-limiting toxicity (DLT) After the observational evaluation period, a decision will be made by the investigator and sponsor based on a discussion of relevant safety data whether to start the next dose group.

SUMMARY:
The goal of this clinical trial is to evaluate the safety and tolerability of multiple doses of human umbilical cord mesenchymal stem cell injection in patients with Ankylosing Spondylitis, and to further explore the efficacy, pharmacodynamic profile and appropriate dose of administration to provide a basis for the use of safer and more effective treatments for patients with Ankylosing Spondylitis in the future.

Participants are required to sign an informed consent form and, after undergoing a series of tests and meeting the protocol's entry and exclusion criteria, are assigned to a dose group for intravenous infusion of human umbilical cord mesenchymal stem cells.

DETAILED DESCRIPTION:
Ankylosing spondylitis (AS) is an inflammatory disease of unknown origin that mainly affects the sacroiliac joints, spinal prominences, paraspinal soft tissues and peripheral joints, and may be accompanied by extra-articular manifestations, and in severe cases, spinal deformities and ankylosis. The etiology of AS is still unclear, but epidemiology shows a strong association with genetic and environmental factors. Treatment is aimed at relieving signs and symptoms, restoring physical function, preventing joint damage, improving quality of life, and preventing complications of spinal disorders. Treatment methods include patient education such as physical exercise and proper posture in life and sleep; pharmacological treatment such as non-steroidal anti-inflammatory drugs (NSAIDs), biologics (e.g. TNF-α antagonists, IL-17 antagonists), DMARDs (e.g. salbutamol, methotrexate), glucocorticoids, etc. In addition, surgical methods such as total hip arthroplasty are also available. Despite these therapeutic or disease control methods, none of them can stop the radiological progression of AS, restore the structural damage of patients, or achieve a cure for the disease.

Stem cells are undifferentiated cells that exist in embryonic or adult tissues and have the potential for self-renewal replication and multidirectional differentiation. Mesenchymal stem cells (MSCs) are one of the most used stem cells in basic and clinical research. According to the literature, MSCs have the ability to migrate and nest in diseased and damaged tissues in vivo, and repair damaged tissues through their multidirectional differentiation potential. MSCs can also improve the local microenvironment, support and promote the regeneration and differentiation of endogenous stem cells, exert anti-inflammatory effects and regulate immunity through their paracrine mechanisms. The collection of human umbilical cord derived mesenchymal stem cells (hUC-MSCs) is non-invasive and there are no medical ethics issues in obtaining them.

There are no medical ethics issues in obtaining them. Similar to other tissue-derived MSCs, hUC-MSCs have a unique self-renewal capacity and multidirectional differentiation potential, such as the ability to differentiate into adipose, bone, cartilage, nerve and liver cells [6]. These properties make hUC-MSCs have the theoretical possibility to treat AS.

Currently, studies on MSCs for the treatment of ankylosing spondylitis (AS) are in the exploratory stage, and several studies have confirmed the safety and efficacy of MSCs for the treatment of AS.

The primary objective of this clinical trial was to examine the safety and tolerability of human umbilical cord MSC injection in patients with AS, and the secondary objective was to examine the initial effectiveness of human umbilical cord MSC injection in treating patients with AS. The trial was designed as a single-arm, single-dose, dose-escalation clinical trial with three dose groups: low-dose group (1,000,000 cells/kg), medium-dose group (3,000,000 cells/kg), and high-dose group (5,000,000 cells/kg). A "3+3" dose escalation design was used, with 3-6 subjects included in each dose group, sequentially from the low to the high dose group. Each subject in the high-dose group was enrolled on a case-by-case basis, and each subject in the high-dose group was allowed to enroll in subsequent subjects only after completing at least 7 days of safety observation after dosing. Each subject received only one corresponding dose.

After all subjects in each trial dose group have completed a 4-week (28-day) dose-limiting toxicity (DLT) observation period, the decision to start the next dose group will be made by the investigator and sponsor after discussion of relevant safety data. Subjects will enter the follow-up period after completing the D28 visit, and the investigator will continue to observe the safety and efficacy of the subjects after dosing.

The investigators continued to monitor the safety and efficacy of the drug after administration. If a subject experiences disease progressiona or requires other treatment (including but not limited to biologics), the investigator will determine whether the subject should be discontinued from the patient risk-benefit perspective and discharged from the group as specified; subjects discharged from the group as determined by the investigator will be followed up as specified for long-term follow-up.

Subjects who have completed the DLT observation period in the previous dose group and have confirmed that the drug is safely tolerated, the investigator and sponsor will agree on whether to proceed to the next dose group. Concurrent enrollment in 2 or more dose groups is not permitted. If during the trial a dose group is observed to meet the termination dose creep criteria, the dose escalation will be terminated and a decision to continue the study with a downward dose adjustment will be made by the investigator and sponsor. The previous dose in the dose group that reached the termination criteria was designated as the maximum tolerated dose (MTD). If the MTD has not been explored and the subject is still safely tolerated after completion of the highest dose group (5,000,000 cells/kg) preset for this trial, the decision to continue with a higher dose escalation will be made by the investigator in consultation with the sponsor.

The extent of adverse events observed in the trial will be determined by the CTCAE 5.0 grading scale, with the following The dose creep will be terminated and the investigator and sponsor will mutually agree whether to use the previous dose as the MTD for the single dose tolerance trial. MTD of the dosing tolerance test.

1. 1 DLT in 3 subjects in a dose group; 3 additional subjects will be included in that dose group for tolerance testing;
2. If ≥2 DLTs occur in 6 subjects in a dose group, the previous dose level of that dose level defined as MTD and dose escalation was stopped.

If the maximum dose group is reached and still no MTD is defined, the investigator and sponsor consult to determine if continued creep.

ELIGIBILITY:
Inclusion Criteria:

* A definitive diagnosis of ankylosing spondylitis (AS) (according to the 1984 New York Revised Criteria, Annex 1) with active AS. Active AS is defined as a Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score of ≥4. Active AS is defined as a Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score of ≥4;
* Received at least 2 non-steroidal anti-inflammatory drugs (NSAIDs) for a total of 4 weeks or more prior to screening. Patients who received at least 2 NSAIDs for a total of 4 weeks or more without significant improvement in symptoms as evaluated by the investigator or who were intolerant; if Patients receiving salazosulfapyridine and/or methotrexate should have been on treatment for at least 3 months or longer and on a stable dose for at least 4 weeks or more prior to enrollment. If the patient is receiving salazosulfapyridine and/or methotrexate, the length of treatment prior to enrollment should be at least 3 months and longer and the stable dose at least 4 weeks and longer;
* If the patient is receiving glucocorticosteroid therapy, stabilization for at least 4 weeks prior to enrollment to a dose equivalent to ≤ 10 mg of prednisone/day;
* Patients and spouses who do not plan to have children within 1 week prior to screening and within 6 months after the end of the trial and who agree to to use effective non-pharmacological contraception during the trial;
* Patients voluntarily signed an informed consent form and were willing to cooperate with the trial process.

Note: CT findings may be accepted if the diagnosis is not clear on x-ray.

Exclusion Criteria:

* Those with complete spinal rigidity;
* Those with hypersensitivity to known components of the test drug, or a history of severe allergy.
* Persons with a history of any malignancy (except basal cell carcinoma of the skin, carcinoma in situ) within 5 years prior to dosing
* Persons with a cardiovascular or cerebrovascular event (heart attack, ischemic or hemorrhagic stroke (except lacunar cerebral infarction), severe cardiac arrhythmia, deep vein thrombosis, etc.) within 3 months prior to dosing
* Those who have had a serious infection or have an active infection requiring intravenous antibiotic treatment within 4 weeks prior to screening
* Lactating females or females with positive blood pregnancy test results at screening/baseline
* Persons with known human immunodeficiency virus infection or impaired immune function or infectious disease (e.g. HBsAg positive, HBcAb positive with HBV-DNA titer > 1000 IU/ml, HCV-Ab, HIV-Ab, syphilis test (TRUST), tuberculosis test (T-SPOT.TB) positive);
* Patients who have participated in other clinical trials or studies within 2 months prior to dosing;
* Those who have been treated with TNF-alpha antagonists or other biological agents within 3 months prior to dosing
* Those who have received DMARDs class drugs within 1 month prior to dosing (except for those treated with salazosulfapyridine or methotrexate for 3 months or more prior to screening and at a stable dose for at least 4 weeks or more) with leflunomide discontinuation <8 weeks; or those with discontinuation time <7 drug half-lives depending on the actual drug class (i.e. DMARDs class drug elution period should exceed 7 half-lives of the corresponding drug), whichever is longer;
* Those whose screening or baseline phase examination meets any of the following: Glutamic aminotransferase (AST) or glutamic alanine aminotransferase (ALT) > 2.5 x ULN (non-hepatic source excluded); Serum creatinine > 1.5 x ULN or glomerular filtration rate a < 60 mL/min/1.73 m2; Activated partial thromboplastin time (APTT) >1.5×ULN or prothrombin time (PT) > 2.5 x ULN (not receiving anticoagulation); Left ventricular ejection fraction ≤ 45%.
* Previously treated with stem cell therapy;
* Subjects with any other irreversible condition or symptom with an expected survival of <3 months
* Those who have undergone spinal or joint surgery within 2 months prior to dosing;
* History of alcoholism, mental illness, drug abuse, or use of any drug within 12 months prior to administration;
* Any other condition that, in the judgment of the investigator, makes them unsuitable for participation in this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-08-30 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Event (AE) | Through study completion, an average of 1 year
  Incidence and severity of any adverse events related to the treatment of the trial drug that occurred during the clinical trial
Maximum tolerated dose (MTD) | Through study completion, an average of 1 year
  Explore the MTD after administration of the test drug

SECONDARY OUTCOMES:
Improvement of Assessment in ankylosingspondylitis 20 (ASAS20) | Baseline, Day 14, Day 28, Week 12, Week 24, Week 36, Week 48
  The ASAS Response Criteria (ASAS 20) is defined as an improvement of at least 20% and an absolute improvement of at least 10 units on a 0-100 scale in at least three of the following domains: Patient global assessment, Pain assessment, Function, and Inflammation.
Improvement of Assessment in ankylosingspondylitis 50 (ASAS50) | Baseline, Day 14, Day 28, Week 12, Week 24, Week 36, Week 48
  The ASAS Response Criteria (ASAS 20) is defined as an improvement of at least 50% and an absolute improvement of at least 10 units on a 0-100 scale in at least three of the following domains: Patient global assessment, Pain assessment, Function, and Inflammation.
Change of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | Baseline, Day 14, Day 28, Week 12, Week 24, Week 36, Week 48
  BASDAI is the most widely used measure of disease activity in axial spinal arthritis (axSpA) and includes the assessment of fatigue, overall low back pain, pain and swelling of peripheral joints, attachment inflammation, severity of morning stiffness discomfort, and duration of morning stiffness. This score is used to compare patients' improvement from baseline. The higher the score is, the more severe the disease is.
Change of Bath Ankylosing Spondylitis Functional Index (BASFI) | Baseline, Day 14, Day 28, Week 12, Week 24, Week 36, Week 48
  BASFI is a scoring measure used to assess the status of their physical function, which relates to the activity performance and functional ability of patients with AS in daily life. This score is used to compare patients' improvement from baseline. The higher the score is, the more severe the disease is.
Change of Bath Ankylosing Spondylitis Metrology Index (BASMI) | Baseline, Day 14, Day 28, Week 12, Week 24, Week 36, Week 48
  BASMI identifies clinically significant changes in spinal movement based on axial (neck, back, lumbar, hip, and pelvic soft tissue) movements in patients with AS. It includes five clinical measures of axial mobility: cervical rotation, tragus to wall distance, lumbar lateral flexion, lumbar flexion, and interankle distance. This score is used to compare patients' improvement from baseline. The higher the score is, the more severe the disease is.
Change of Ankylosing Spondylitis Disease Activity Score (ASDAS) | Baseline, Day 14, Day 28, Week 12, Week 24, Week 36, Week 48
  ASDAS is a new comprehensive index for evaluating AS disease activity, which includes 5 questions:
  Q1: Overall low back pain level; Q2: Overall patient evaluation: How would you describe your average disease activity over the past week? Score 0-10, 0 is inactive, 10 is very active; Q3: Pain and swelling degree of peripheral joints; Q4: Morning stiffness duration; Q5: Acute phase reactants: C-reactive protein level (CRP, mg/L) or erythrocyte sedimentation rate level (ESR, mm/h)
Change of Patient's global assessment of disease activity (PtGADA) | Baseline, Day 14, Day 28, Week 12, Week 24, Week 36, Week 48
  Patients were asked questions about how affected they were by the disease and were evaluated using a 0-10 rating scale, with higher scores indicating worse disease status.
Physician's global assessment of disease activity (PhGADA) | Baseline, Day 14, Day 28, Week 12, Week 24, Week 36, Week 48
  The question of the extent to which the patient is affected by the disease is assessed by the doctor and evaluated using a 0-10 scoring scale, with the higher the score indicating the worse the disease status.
Modified stoke ankylosing spondylitis spinal score (mSASSS) | Baseline, Week 48
  SASSS scores are based on the presence of erosion, hardening, squaring of the posterior and anterior corners of the lumbar spine, osteophytes formation, and whole bone bridging, and are less sensitive to change. mSASSS adds a score to the cervical spine on the basis of SASSS, ranging from 0 to 72 points. A higher score indicates a higher severity of the patient's disease.
Ankylosing Spondylitis spine Magnetic Resonance Imaging-activity (ASspiMRI) | Baseline, Week 48
  ASspiMRI is the first MRI scoring system to evaluate changes in spinal inflammation in patients with AS. The scoring system requires a semi-quantitative analysis of at least two images/lesion areas for all accessible vertebrae (C2-S1, n=23), intervertebral Spaces, and intervertebral discs. A higher score indicates a higher severity of the patient's disease.
Erythrocyte sedimentation Rate (ESR) | Baseline, Day 2, Day 3, Day 7, Day 14, Day 28, Week 12, Week 24, Week 36, Week 48
  To explore the rate of erythrocyte sedimentation. ESR can also help to observe the changes of the disease, the rate of ESR is accelerated in the active period, and the rate of ESR is slowed down when the disease is improved. The inactive ESR can be restored to the reference range.
C-reactive protein (CRP) | Baseline, Day 2, Day 3, Day 7, Day 14, Day 28, Week 12, Week 24, Week 36, Week 48
  To explore the concentration of C-reactive protein. CRP is closely related to other inflammatory factors such as erythrocyte sedimentation rate, which can reflect the inflammation in patients.

OTHER OUTCOMES:
Interleukin-2 (IL-2) | Baseline, Day 2, Day 3, Day 7, Day 14, Day 28, Week 12, Week 24, Week 36, Week 48
  The concentration of IL-2
Interleukin-6 (IL-6) | Baseline, Day 2, Day 3, Day 7, Day 14, Day 28, Week 12, Week 24, Week 36, Week 48
  The concentration of IL-6
Interleukin-17 (IL-17) | Baseline, Day 2, Day 3, Day 7, Day 14, Day 28, Week 12, Week 24, Week 36, Week 48
  The concentration of IL-17
Interleukin-22 (IL-22) | Baseline, Day 2, Day 3, Day 7, Day 14, Day 28, Week 12, Week 24, Week 36, Week 48
  The concentration of IL-22
Interleukin-23 (IL-23) | Baseline, Day 2, Day 3, Day 7, Day 14, Day 28, Week 12, Week 24, Week 36, Week 48
  The concentration of IL-23
Tumor necrosis factor-α (TNF-α） | Baseline, Day 2, Day 3, Day 7, Day 14, Day 28, Week 12, Week 24, Week 36, Week 48
  The concentration of TNF-α
Transforming growth factor-β (TGF-β） | Baseline, Day 2, Day 3, Day 7, Day 14, Day 28, Week 12, Week 24, Week 36, Week 48
  The concentration of TGF-β
Interferon-γ (IFN-γ) | Baseline, Day 2, Day 3, Day 7, Day 14, Day 28, Week 12, Week 24, Week 36, Week 48
  The concentration of IFN-γ
Monocyte chemotactic protein [MCP]-1 (CCL-2) | Baseline, Day 2, Day 3, Day 7, Day 14, Day 28, Week 12, Week 24, Week 36, Week 48
  The concentration of CCL-2
Helper T cell 1 (Th1) | Baseline, Day 2, Day 3, Day 7, Day 14, Day 28, Week 12, Week 24, Week 36, Week 48
  The concentration of Th1
Helper T cell 2 (Th2) | Baseline, Day 2, Day 3, Day 7, Day 14, Day 28, Week 12, Week 24, Week 36, Week 48
  The concentration of Th2
Regulatory T cells (Treg) | Baseline, Day 2, Day 3, Day 7, Day 14, Day 28, Week 12, Week 24, Week 36, Week 48
  The concentration of Treg
Helper T cell 17 (Th17) | Baseline, Day 2, Day 3, Day 7, Day 14, Day 28, Week 12, Week 24, Week 36, Week 48
  The concentration of Th17
Cluster of differentiation 3+ (CD3+) | Baseline, Day 2, Day 3, Day 7, Day 14, Day 28, Week 12, Week 24, Week 36, Week 48
  The concentration of CD3+
Cluster of differentiation 4+ (CD4+) | Baseline, Day 2, Day 3, Day 7, Day 14, Day 28, Week 12, Week 24, Week 36, Week 48
  The concentration of CD4+
Cluster of differentiation 8+ (CD8+) | Baseline, Day 2, Day 3, Day 7, Day 14, Day 28, Week 12, Week 24, Week 36, Week 48
  The concentration of CD8+
Cluster of differentiation 4+ / Cluster of differentiation 8+ (CD4+/CD8+) | Baseline, Day 2, Day 3, Day 7, Day 14, Day 28, Week 12, Week 24, Week 36, Week 48
  The ratio of CD4+/CD8+
Immunoglobulin A (IgA) | Baseline, Day 2, Day 3, Day 7, Day 14, Day 28, Week 12, Week 24, Week 36, Week 48
  The concentration of IgA
Immunoglobulin G (IgG) | Baseline, Day 2, Day 3, Day 7, Day 14, Day 28, Week 12, Week 24, Week 36, Week 48
  The concentration of IgG
Immunoglobulin M (IgM) | Baseline, Day 2, Day 3, Day 7, Day 14, Day 28, Week 12, Week 24, Week 36, Week 48
  The concentration of IgM

CONTACTS AND LOCATIONS:
Overall Officials: Chunde Bao, Principal Investigator — RenJi Hospital

IPD SHARING:
Plan to Share IPD: No